CLINICAL TRIAL: NCT06499363
Title: Treprostinil in Newborns With Pulmonary Hypertension; a Noninterventional Study to Collect Data on Drug Utilization, Safety, and Effectiveness.
Brief Title: Treprostinil in Newborns With Pulmonary Hypertension; a Non-Interventional Study to Collect Data on Drug Utilization, Safety, and Effectiveness
Acronym: NEPHY
Status: Recruiting | Type: Observational
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: FREM-NIS-2301
Record Dates: First submitted 2024-05-21; First posted 2024-07-12 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Persistent Pulmonary Hypertension of Newborn
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study will seek to describe the uses and safety and efficacy outcomes of treprostinil in clinical practice in patients with persistent pulmonary hypertension (PPHN).

ELIGIBILITY:
Inclusion Criteria:

1. Newborn infants who received at least one dose of IV or SC treprostinil as per clinical practice within 5 years from the moment of data collection.
2. Aged up to 44 weeks after conception at treprostinil initiation.
3. Pulmonary hypertension (PH) or suspicion of PH at the moment of treprostinil initiation.
4. Parent(s) or legally authorized representative(s) provides non-opposition consent for the patient participation in the study.
5. Newborn infants affiliated to French social security.

Exclusion Criteria:

* None.

Max Age: 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Approximately 60 newborns with PH (of whom at least 40 newborns with persistent pulmonary hypertension of the newborn [PPHN]) are expected to be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Characteristics of neonates receiving treprostinil in the clinical practice. | From baseline to Day 30 after last dose of treprostinil
  Sex (male/female) ; Gestational Age (weeks) ; Birth Weight (g) ; Apgar (1 and 5 min, 0-10) and Time from birth to treprostinil initiation (h)
Treprostinil-specific treatment patterns. | From baseline to Day 30 after last dose of treprostinil
  Prior concomitant treatments, treprostinil route, treprostinil dose(s) (mg/ml) and treprostinil treatment duration (days).
Number of participants with treatment-related adverse events to evaluate safety. | From baseline to Day 30 after last dose of treprostinil

SECONDARY OUTCOMES:
Composite endpoint of absence of complications through Day 14 after the index date. | From baseline to Day 30 after last dose of treprostinil
Description of the clinical outcomes from treprostinil start day (i.e., Day 0) to Day 14 and at Day 30 after last dose of treprostinil. | 0h, 24h, 48h, 72h, Day 7, Day 14, and Day 30 after last dose of treprostinil (if applicable).
  Evolution of pre- and post-ductal oxygen saturation (SpO2); oxygen partial pressure (PO2); clinical laboratory parameters and fraction of inspired oxygen (FiO2) at times 0h, 24h, 48h, 72h, Day 7, Day 14, and Day 30 after last dose of treprostinil.
Description of neurodevelopmental progress over 2 years after treprostinil initiation through a Global Clinical Impression Scale. | From day 30 after treprostinil treatment to Year 2 after last dose of treprostinil

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Lyon (HCL) - Hopital Femme Mère Enfant, Bron
  - Réanimation néonatale CHU Grenoble Alpes - Hôpital Couple Enfant, Grenoble
  - CHU Lille - Clinique de Néonatalogie, Lille
  - CHU de Toulouse Hopital des enfants - Réanimation Néonatale, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided